CLINICAL TRIAL: NCT04814706
Title: Ultrasound Assessment of Gastric Volume in Elderly Patients Undergoing Staged-bilateral Total Knee Arthroplasty After Drinking Carbohydrate-containing Fluids: A Prospective Observational Comparative Study
Brief Title: Gastric Volume in Elderly Patients Undergoing Staged Bilateral Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2103/673-302
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Arthritis Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group C: Patients drank carbohydrate fluid 2 hours prior to surgery.
  Interventions: Dietary Supplement: Carbohydrate drinking

INTERVENTIONS:
Dietary Supplement: Carbohydrate drinking — Administration of carbohydrate fluid

SUMMARY:
In the past, some guidelines advised no oral intake for at least 8 hours before any surgery, However, research has shown risks associated with excessive fasting, such as postoperative insulin resistance, and advantages in shorter fasting protocols, such as reduced postoperative nausea and vomiting.

The perioperative fasting guidelines of the European Society of Anaesthesiology focus on preoperative carbohydrates. They hold that it is safe for patients to drink carbohydrate-rich fluids up to 2 hours before elective surgery and that drinking carbohydrate-rich fluids improves subjective well-being, reduces thirst and hunger, and reduces postoperative insulin resistance at an evidence level of 1++. Nevertheless, data on drinking carbohydrate fluids before surgery in elderly patients are limited.

Some factors have been known to influence the gastric emptying rate, as for example, old age, pain, and the use of opioid analgesics.

In the previous study, evidence of increased pain was reported in patients undergoing staged bilateral total knee arthroplasty, in whom the second operated knee had greater sensitivity (tertiary hyperalgesia) due to the surgical injury to the first operated knee.

In the present study, the investigators will evaluate the effect of old age, surgical stress, pain, and the use of analgesics on the residual gastric volume in elderly patients undergoing staged-bilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for staged bilateral total knee arthroplasty aged 65 to 85 years
* American Society of Anesthesiologists physical status classification 1, 2, and 3
* Body mass index < 35 kg/cm2
* Patients administered carbohydrate-containing fluid 2 hours prior to surgery

Exclusion Criteria:

* Previous surgery of the upper gastrointestinal tract
* Achalasia
* Diabetes

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Study Population: Study participants will be patients whom are scheduled to undergo staged bilateral total knee arthroplasty requiring administration of carbohydrate-containing fluid 2 hours prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Gastric volume 1 | First stage operation, during the gastric volume measuring at preoperative holding area/ an average of 30 minutes
  Gastric volume measured before induction of spinal anesthesia using ultrasound
Gastric volume 2 | Second stage operative, during the gastric volume measuring at preoperative holding area/ an average of 30 minutes
  Gastric volume measured before induction of spinal anesthesia using ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea